CLINICAL TRIAL: NCT00611494
Title: A Single Centre, Prospective, Open-Label, Parallel Group, Randomized Study to Compare the Gastrointestinal Tolerability of Mycophenolate Mofetil (MMF, CellCept) and Enteric-Coated Mycophenolate Sodium (EC-MPS, Myfortic) in Maintenance Transplant Patients Treated With Calcineurin Inhibitors
Brief Title: Gastrointestinal Tolerability of MMF vs EC-MPS in Maintenance Transplant Patients Treated With Calcineurin Inhibitors
Acronym: MOTOR-MPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. George Therapondos, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0398-A
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Organ Transplantation
Keywords: Drug tolerance; Quality of Life
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): MMF
  Interventions: Drug: MMF
- B (Active Comparator): EC-MPS
  Interventions: Drug: EC-MPS

INTERVENTIONS:
Drug: MMF — Gradual optimization of drug dosage, as clinically tolerated.
  Other Names: CellCept
  Arms: A
Drug: EC-MPS — Conversion from MMF to EC-MPS. Gradual optimization of drug dosage, as clinically tolerated.
  Other Names: Myfortic
  Arms: B

SUMMARY:
The purpose of the study is to assess the gastrointestinal tolerability of EC-MPS compared to MMF in maintenance transplant patients on a calcineurin inhibitor regimen, who require MMF dose reductions of 25% or more due to GI complications. The tested hypothesis is that the EC-MPS treatment is superior to the MMF therapy in terms of tolerability and that patients on the EC-MPS formulation will be able to tolerate higher doses compared to those on MMF.

DETAILED DESCRIPTION:
The use of mycophenolate mofetil (MMF) in combination with a calcineurin inhibitor (CNI: tacrolimus or cyclosporine) has been shown to improve graft survival in renal, cardiac and liver transplantation patients. However, its use has been associated with significant side effects, including gastrointestinal complications, causing dose reductions, interruption or termination of the therapy. An alternate formulation: enteric coated mycophenolate sodium (EC-MPS) was designed to alleviate the severity of upper gastrointestinal side effects. Several trials detailed in the protocol suggest a benefit in GI related health following conversion from MMF to EC-MPS, however we believe that robust data are lacking.

ELIGIBILITY:
Inclusion Criteria:

* recipients of liver or kidney or heart or lung or kidney/pancreas transplants
* at least 1 month post solid organ transplant
* on an immunosuppressive regimen which includes MMF in combination with cyclosporine A or tacrolimus
* previous MMF dose reduction of minimum of 25% of total dose due to at least one gastrointestinal complication with MMF therapy
* age of 18-75 years

Exclusion Criteria:

* less than 1 month post transplant
* allergy (hypersensitivity) to MPA, MMF, EC-MPS or to any ingredients of Myfortic or CellCept
* unwillingness or inability to give written consent
* pregnant or nursing women, or women planning to become pregnant
* patients with GI symptoms due to reasons other than related to MMF therapy
* active Post Transplant Lymphoproliferative Disease (PTLD)
* significant or uncontrolled concomitant infections or other serious medical problems
* active bacterial, viral or fungal infection
* inability to self-administer the Quality of Life questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The number of patients with at least 1 GI symptom that is continuing or starting after the 1-month dose stabilization period | 12 months

SECONDARY OUTCOMES:
Analysis and comparison of various Gastrointestinal Symptom Rating and Quality of Life Questionnaire (the GSRS, GIQLI, PGWB,OTE for HRQoL) scores across and within the 2 cohorts. | At months 1, 3, 6, 12 post-study start
Incidence and severity of adverse events | months 3, 6, 12
Patient survival, graft survival and rejection episodes across the 2 cohorts | months 3, 6, 12
Dose reductions, interruptions, fractionations and patient withdrawals across the two cohorts due to adverse events | Months 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: George Therapondos, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital - Multi Organ Transplant Program, Toronto, Ontario, Canada